CLINICAL TRIAL: NCT06432387
Title: Coagulation Factors Alterations in Patients Undergoing Complex Thoraco-abdominal Aortic Aneurysm Repair (CoFA-TAAA); a Prospective Observational Study
Brief Title: Coagulation Factors Alterations in Patients Undergoing Complex Thoraco-abdominal Aortic Aneurysm Repair
Acronym: CoFA-TAAA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anaesthesiology, University of Thessaly
Other Study IDs: CoFA-TAAA
Record Dates: First submitted 2024-05-08; First posted 2024-05-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Thoraco-abdominal Aortic Aneurysm Repair; Coagulation Factors Alterations; Platelet Activation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing complex thoraco-abdominal aortic aneurysm repair: Perioperative laboratory examinations will follow institutional guidelines. These will include, but will not be limited to full blood count, conventional coagulation tests, liver function, and kidney function tests. Moreover, for the purpose of this study, the following parameters will also be obtained; vWF, factors VIII and XI, D-dimers, fibrinogen, platelets activation (multiplate), adams-13, anti-Xa and high sensitivity troponin. All samples will be obtained via puncture from a peripheral vein. Blood samples will obtained at three time points; preoperatively before induction to GA (01), postoperative day 1 (02) and postoperative day 3rd-4th (03). During hospitalization any myocardial injury after non cardiac surgery, acute kidney injure and post-implantation syndrome will be recorded.
  Of note, at 30 days, 3, 6 and 12 months our patients will undergo an evaluation for any major cardiovascular event, implant failure or death of any cause.
  Interventions: Other: Patients undergoing complex thoraco-abdominal aortic aneurysm repair

INTERVENTIONS:
Other: Patients undergoing complex thoraco-abdominal aortic aneurysm repair — Patients undergoing complex thoraco-abdominal aortic aneurysm repair

SUMMARY:
This study will evaluate the impact of complex thoraco-abdominal aortic aneurysm repair in coagulation during the immediate postoperative period in patients undergoing omplex thoraco-abdominal aortic aneurysm repair.

DETAILED DESCRIPTION:
Endovascular aneurysm repair of abdominal aorta activates a significant inflammation reaction and has an impact on coagulation. Platelet activation seems to have a major role in this prothrombotic and hypercoagulable state. In complex thoraco-abdominal aortic aneurysm repair the implants are more complexed and the duration of operation longer. The main hypothesis is that all the above have a greater impact on platelet activation and coagulation alterations.

The aim of this study is the evaluation of the impact of complex thoraco-abdominal aortic aneurysm repair in coagulation during the immediate postoperative period in patients undergoing omplex thoraco-abdominal aortic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing complex thoraco-abdominal aortic aneurysm repair in University Hospital of Larissa, after informed consent will be included.

Exclusion Criteria:

* Refuse to participate
* Prior surgery within 3 months
* ASA PS > 3
* Known medical history of thrombophilia or functional platelet dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be treated by the same medical team in UHL according to the European Society for Vascular Surgery (ESVS) guidelines. Preoperatively patients will be treated with aspirin 100 mg once daily for at least 5 days. Postoperatively in the absence of bleeding patients will receive aspirin 100 mg and in the absence of neurological dysfunction due to spine ischemia they will receive clopidogrel 150 mg and from the next day dual antiplatelet therapy (aspirin 100 mg and clopidogrel 75 mg). If the patient was treated with anticoagulant agents this will be discontinued preoperative according to ACCP guidelines and it will be restarted on the 1st or 2nd postoperative day based on hemostasis. In this case patients will be treated with aspirin 100 mg once daily five days preoperatively and aspirin will also be continued postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Coagulation status | Day of surgery, 1st postoperative day, 4-5th postoperative day
  Early preoperatively, early and late postoperatively
Myocardial injury after non cardiac surgery | Day of surgery, 1st postoperative day, 4-5th postoperative day
  Early preoperatively, early and late postoperatively
Acute kidney injury | Day of surgery, 1st postoperative day, 4-5th postoperative day
  Early preoperatively, early and late postoperatively
Post-implantation syndrome | Day of surgery, 1st postoperative day, 4-5th postoperative day
  Early preoperatively, early and late postoperatively
Major cardiovascular events | Day of surgery, 1st postoperative day, 4-5th postoperative day
  Early preoperatively, early and late postoperatively
Major cardiovascular events, implant failure and death of any cause | 30 days, 3, 6, and 12 months postoperatively
  Early preoperatively, early and late postoperatively and 1 at one month

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, Prof, Study Chair — University of Thessaly
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No